CLINICAL TRIAL: NCT00410345
Title: Cervical Rippening With Antiprogesterone in Midtrimester Abortions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mifepristoneoxytocin-HMO-CTIL
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2008-05

CONDITIONS: Abortion, Missed
MeSH Terms: conditions — Abortion, Missed | interventions — Mifepristone

ARMS (2):
- Pitocin (Experimental): Treatment with Pitocin after mifegine
  Interventions: Drug: Mifepristone
- Cytotec (Active Comparator): Treatment with cytotec after mifegine
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone

SUMMARY:
Induction of midtrimester abortion includes cervical ripening and then contraction to induce uterine evacuation. There are several protocols, but most of them include using prostaglandins (PG). The disadvantages of using PG include uncomfortable side effects and limits of using it for women after cesarean section. Mifepristone is an antiprogesterone drug and been used for induction of abortion in first and second trimesters abortions. The aim of this study is to explore the effectiveness of Mifepristone for cervical ripening before high dose Oxytocin drip.

DETAILED DESCRIPTION:
The aim of this study is to explore the effectiveness of Mifepristone for cervical ripening before high dose Oxytocin drip in midtrimester abortions. After informed consent, all the women will be randomized for Mifepristone or placebo. 48 hours later, high dose oxytocin drip will be started and we will examine the success rate to induce abortion, the duration from starting oxytocin till evacuation of uterus and side effects.

ELIGIBILITY:
Inclusion Criteria:

* midtrimester late abortion
* midtrimester induced abortion

Exclusion Criteria:

* placenta previa
* infected abortion
* rupture of membranes
* s/p cesarean section *2 or more

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2004-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
success of abortion induction
abortion induction duration

CONTACTS AND LOCATIONS:
Overall Officials: Assaf Ben-Meir, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel